CLINICAL TRIAL: NCT02894450
Title: Study of Clinical and Laboratory Variables Associated With a Direct Oral Anticoagulant Bioassay (Xaban) Higher Among Those Aged Over 75 Years, as AOD for Atrial Fibrillation
Brief Title: Study of Clinical and Laboratory Variables Associated With a Direct Oral Anticoagulant Bioassay Higher Among Those Aged Over 75 Years
Acronym: AOD-SA
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0402
Record Dates: First submitted 2016-08-11; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; oral anticoagulant; bioassay; elderly subject
MeSH Terms: conditions — Atrial Fibrillation | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: blood test — bioassay xaban

SUMMARY:
The objective of this study was to investigate whether there is a link between clinical and biological variables and bioassay high xaban in elderly patients as part of an unscheduled hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 75 years
* Entering SAU or MPG (Nantes University Hospital) as part of an unscheduled hospitalization for acute or subacute disease (About MPG, will be included patients admitted to the department within 48 hours of calling the doctor)
* In xaban to entry (dabigatran, rivaroxaban, Apixaban) for non-valvular atrial fibrillation
* In whom hemostasis tests will be prescribed as part of usual care
* Patient has given its verbal agreement

Exclusion criteria

Patients with the following criteria may not be included:

* Patients refusing to participate in the study
* Patients under guardianship
* Inability to obtain the date and time of the last dose of xaban

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients over 75 years under anticoagulant treatment 'xaban' (dabigatran, rivaroxaban, Apixaban) for atrial fibrillation, hospital unscheduled manner in Medicine and Geriatric services Versatile Service Home Emergency CHU Nantes and where a hemostatic balance is expected to be offered the study.
  The recruitment will be made on a 6-month period (November 2014 - April 2015). Bioassay 'xaban' will be made from the remainder of the tube removed for hemostasis tests provided in the usual care of patients.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
bioassay direct oral anticoagulants | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Chevalet, Dr, Principal Investigator — Nantes University Hospital